CLINICAL TRIAL: NCT06534294
Title: Effect of Non-pharmacological Anti-anxiety Exercises on Perceived Stress and Cortisol Level Before Elective Per Cutaneous Transluminal Coronary Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Afify, Associate professor, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IHC00070
Record Dates: First submitted 2024-07-15; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty
MeSH Terms: interventions — Musculoskeletal Manipulations; Breathing Exercises; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP1 (Experimental): Reflexology procedure will applied to patients in calm, quiet patient room with adequate light and in the supine position. For the relaxation of patients 10 minutes of relaxation techniques and stimulation of the reflexology points before reflexology, Reflex therapy was done for each patient for 30 minutes, first for the right foot and then for the left foot (15 minutes each)
  Interventions: Other: reflexology
- GROUP2 (Experimental): patients carried out breathing exercises AS 3 stages(13), stage one Beginning stage for 5 minutes will ask the patients to Sit , Flatten the shoulders, open the legs, and place your arms at your sides naturally , Close eyes and focus on present feelings , stage two deep breathing stage for 10 minutes Exercises were deep breathing exercises; deep inspiration for 5 seconds and slow prolonged expiration for next 5 seconds, at a rate of 6 breaths/min, rest for one minute after each cycle , then apply the exercises again , end stage ; Close eyes and focus your present feelings, Then Relax the whole body for 5 minutes.
  Interventions: Other: breathing exercise
- GROUP3 (Experimental): procedure that will done in reflexology and deep breathing will applied
  Interventions: Other: reflexology; Other: breathing exercise
- GROUP4 (Other): In this group: will received only standard care
  Interventions: Other: standard care

INTERVENTIONS:
Other: reflexology — Reflex therapy was done for each patient for 30 minutes, first for the right foot and then for the left foot (15 minutes each) and breathing exercises in 3 stages
  Arms: GROUP1; GROUP3
Other: breathing exercise — breathing exercise done as 3 stages,stage one for 5 minutes, stage two for 10 minutes end stage ; Close eyes and focus your present feelings, Then Relax the whole body for 5 minutes.
  Arms: GROUP2; GROUP3
Other: standard care — standard medical care no other treatment
  Arms: GROUP4

SUMMARY:
Effect of non-pharmacological anti-anxiety exercises on Perceived Stress and cortisol level before elective percutaneous transluminal coronary angioplasty

DETAILED DESCRIPTION:
patients will be selected from national heart institute their age from 30 -50 years old. Patients will be assigned randomly into 4 groups 15 in each group, reflexology group, deep breathing group, combined group (reflexology and deep breathing) and control group. Before procedure two tools will used to collect data (demographic characteristics format the beginning once and Distress Thermometer scale before and 30 minutes after application in all groups ) in addition blood samples (5 mL) will take from all the patients on an empty stomach between 08:30 and 10:00 in the morning and 30 minutes after the application to determine the cortisol level in all groups

ELIGIBILITY:
Inclusion Criteria:

* Fully conscious patients, aged from 30 to 50 years.
* will do percutaneous transluminal coronary angioplasty for the first time without any problem of communication.
* accepting to give Blood samples available between 08:30 and 10:00 in the morning (to avoid differences in cortisol levels), and agreeing to participate in the study

Exclusion Criteria:

* having myocardial infarction symptoms,
* unconscious, having a surgery in the last 6 weeks,
* previously diagnosed with a psychiatric disorder or still having a psychiatric disease, using anxiety medication (psychotropic), corticosteroid, using estrogen or amphetamine derivative drugs,
* infection of the lower extremities, having varicose veins, having peripheral neuropathy and deep vein thrombosis or risk of development, high fever,

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Cortisol Levels | At subject enrollment "single session"
  2 tubes of blood samples (5 mL) will take from the patients in all groups on an empty stomach between 08:30 and 10:00 in the morning and 30 minutes after the application to determine the cortisol level
Distress Thermometer | At subject enrollment "single session"
  It is a visual analog scale consisting of only 1 question that patients can apply on their own. On the scale, there is a thermometer with numbers from 0 to 10. A score of 0 indicates that the individual has no distress, and a score of 10 indicates distress at the highest limit.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menofia, Egypt